CLINICAL TRIAL: NCT01994421
Title: Effects of Kinesiotape on Quadriceps and Hamstring Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Amar Arhab, Mr, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: UGeneva
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Facilitating kinesiotape; Inhibiting kinesiotape; Classical tape; No tape
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (1):
- Kinesiotape (Sham Comparator)
  Interventions: Other: Kinesiotape

INTERVENTIONS:
Other: Kinesiotape

SUMMARY:
Background: Kinesiotaping (KT) is an elastic therapeutic tape developed in the 70's by Dr Kenso Kase for prevention and treatment of sports injuries. Research shows that through activation of skin receptors KT improves blood and lymph flow, increases proprioception, helps relieve pain, facilitates joint and muscle alignment, and enhances muscle function. Despite the increasing popularity of KT, uncertainty remains regarding, in particular, its effectiveness in improving strength.

Purpose: The purpose of the current study was to investigate the short-term effects of KT on muscle strength when applied to the quadriceps muscles of healthy subjects.

Methods: A randomized controlled trial with 52 healthy subjects was conducted. Subjects were tested under four different conditions: a) facilitating Kinesiotape, b) inhibiting Kinesiotape, c) classical tape with no elastic properties, and d) no-taping across four different sessions. The parameters of interest were: quadriceps and hamstrings maximal strength and power using vertical jump tests (squat jump and countermovement jump), and peak concentric and eccentric knee torque (using isokinetic test protocol).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* allowed to perform jumps

Exclusion Criteria:

* pregnancy
* history of cardio-vascular disease
* antecedents of lower extremity injuries
* use of any doping substances listed by the World Anti-doping Agency
* any contraindication to exercise

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Vertical jump height change with different tapes | Week 1, week 2, week 3, and week 4

SECONDARY OUTCOMES:
Isokinetic knee strength change with different tapes | Week 1, week 2, week 3, and week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Unite d'orthopédie et traumatologie du sport, Geneva, Canton of Geneva, Switzerland